CLINICAL TRIAL: NCT03228992
Title: A DOUBLE-BLIND, REPEAT-DOSE, PARALLEL GROUP, PILOT STUDY COMPARING THE EFFICACY AND SAFETY OF ORALLY ADMINISTERED IBUPROFEN AND PLACEBO IN DELAYED ONSET MUSCLE SORENESS
Brief Title: Ibuprofen Versus Placebo For Muscle Soreness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jean Brown Research (Other)
Responsible Party: Principal Investigator, Derek Muse, Principal Investigator, Jean Brown Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JBR-002
Record Dates: First submitted 2017-05-16; First posted 2017-07-25 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-07

CONDITIONS: Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Active Comparator): Subjects will receive a total of 4 doses of oral ibuprofen 400 mg over a 24 hour period.
  Interventions: Drug: Ibuprofen 400 mg
- Placebo (Placebo Comparator): Subjects will receive a total of 4 doses of oral placebo over a 24 hour period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Subjects will receive 4 doses of oral ibuprofen over a 24 hour period.
  Arms: Ibuprofen
Other: Placebo — Subjects will receive 4 doses of placebo over a 24 hour period.
  Arms: Placebo

SUMMARY:
The study will assess the sensitivity of the Delayed Onset Muscle Soreness Model by comparing the safety and efficacy of oral ibuprofen to placebo over 24 hours.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo controlled, parallel group, pilot safety and efficacy study. Healthy male or female subjects who have a history of occasional muscle soreness and are not currently exercising will be asked to volunteer for the study. All subjects will complete an informed consent process prior to study procedures.

The study duration is anticipated to be approximately 4 months. Each subject may be in the study for up to 45 days including screening, run-in, inpatient and outpatient dosing and assessments, follow-up visit and follow-up telephone contact.

ELIGIBILITY:
Subjects must meet the following criteria to be included in the study:

1. Male or female subjects aged 18-55 years;
2. In good general health;
3. Non-pregnant, non-lactating female subjects must be:

   1. physically incapable of childbearing potential (postmenopausal for more than 1 year or surgically sterile) or
   2. practicing an acceptable method of contraception (hormonal, barrier with spermicide, intrauterine device, vasectomized or same sex partner, or abstinence). Subjects using hormonal birth control must have been on a stable dose of treatment for at least 30 days and received at least 1 cycle of treatment prior to randomization.
4. History of experiencing muscle pain/soreness after moderately strenuous exercise;

Subjects are excluded from the study if any of the following criteria apply:

1. Currently participating in an exercise regimen.
2. Have an allergy or intolerance to any NSAID, aspirin, acetaminophen or lactose;
3. History of rhabdomyolysis;
4. Have participated in an investigational study within the past 30 days of screening;
5. Are an employee or relative of an employee of the study site (directly involved with the study).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Model Sensitivity | 24 hours
  Assess whether ibuprofen provides more relief than placebo in the DOMS model.

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company Website — http://jeanbrownresearch.com